CLINICAL TRIAL: NCT01163552
Title: Surgical Cytoreduction Followed by Intraoperative Intrathoracic Hyperthermic Chemotherapy Perfusion for the Management of Disseminated Pleural Malignancies
Brief Title: Heated Chemotherapy for Cancers That Have Spread to the Chest Cavity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Principal Investigator, Gary Schwartz, MD, St. Luke's-Roosevelt Hospital Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLR IRB#09-207
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Pleural Metastases; Breast Cancer; Colon Cancer; Ovarian Cancer; Uterine Cancer; Renal Cell Cancer; Thymic Cancer
Keywords: pleural metastases
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Carcinoma, Renal Cell; Thymus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical Debulking and Intrathoracic Hyperthermic Chemotherapy (Experimental): Patients in this trial will undergo surgical debulking followed by intrathoracic hyperthermic chemotherapy perfusion.
  Interventions: Procedure: Surgical debulking and Intrathoracic Hyperthermic Chemotherapy

INTERVENTIONS:
Procedure: Surgical debulking and Intrathoracic Hyperthermic Chemotherapy — Surgical debulking of intrathoracic metastases will be performed, followed by perfusion of the chest with heated Cisplatin for 60 minutes.

SUMMARY:
Cancers that have spread to the inner lining of the chest are classified as Stage IV and bear a poor prognosis. Surgery is rarely an option, with palliative chemotherapy and/or radiation therapy the only treatment options. This study intends to evaluate whether surgical removal of all visible tumor on the chest wall followed by bathing the chest cavity in heated chemotherapy solution will improve outcomes for these advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-75 years
2. Radiographic evidence of pleural dissemination with histologically or cytologically confirmed diagnosis.
3. Primary source control (breast, ovarian, uterine, colon, renal cell, thymic cancer)
4. Adequate liver and renal function defined as a bilirubin of < 2.0 mg/dl, albumin > 3.0g/dl, and a creatinine of < 1.5 mg/dl, respectively.
5. Absolute neutrophil count (ANC) of ≥1,500/mm3 and a platelet count ≥100,000/mm3.
6. A Karnofsky Performance Status score of ≥60

Exclusion Criteria:

1. Patients without satisfactory oncological control of their primary cancer.
2. Radiographic evidence of abdominal, pelvic, or intracranial metastatic disease.
3. Chemotherapy and/or radiotherapy must have been completed at least one month prior to entry in the study. Patients may not receive concurrent chemotherapy, immunotherapy, radiotherapy, or any investigational drugs while participating in this study.
4. Significant active medical disease including, but not limited to:

   * Cardiac disease, including: congestive heart failure or angina pectoris; recent (within 1 year) history of a myocardial infarction; uncontrolled hypertension; arrhythmias.
   * Active infections
   * Uncontrolled diabetes mellitus
   * Chronic renal insufficiency
   * HIV/AIDS - routine HIV testing will not be performed, but patients known to be HIV positive will be excluded.
5. Pregnant or lactating women.
6. Allergy to intravenous contrast

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | 1 year
  Most cancers that have spread to the chest cavity have limited survival. Response to systemic chemotherapy and radiation therapy is short-lived. This end point will determine the time to disease progression of this experimental treatment modality.
Survival | 1 year
  Most cancers that have spread to the chest cavity have limited survival. Response to systemic chemotherapy and radiation therapy is short-lived. This end point will determine the overall survival period following treatment with this experimental modality.

SECONDARY OUTCOMES:
Systemic drug absorption | 1 month
  By perfusing the chest cavity with chemotherapy, higher doses can be safely administered as less drug is absorbed systemically and therefore toxicity should be lower. This end point will assess drug toxicity due to intrathoracic perfusion.
Complications | 1 month
  Patients will undergo surgical debulking prior to intrathoracic chemotherapy perfusion. Complications from the surgery as well as inhibited wound healing from chemotherapy will be monitored as a secondary end point.

CONTACTS AND LOCATIONS:
Overall Officials: Cliff P Connery, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center, Division of Thoracic Surgery
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Background] Matsuzaki Y, Shibata K, Yoshioka M, Inoue M, Sekiya R, Onitsuka T, Iwamoto I, Koga Y. Intrapleural perfusion hyperthermo-chemotherapy for malignant pleural dissemination and effusion. Ann Thorac Surg. 1995 Jan;59(1):127-31. doi: 10.1016/0003-4975(94)00614-D. PMID 7818311
- [Background] Ratto GB, Civalleri D, Esposito M, Spessa E, Alloisio A, De Cian F, Vannozzi MO. Pleural space perfusion with cisplatin in the multimodality treatment of malignant mesothelioma: a feasibility and pharmacokinetic study. J Thorac Cardiovasc Surg. 1999 Apr;117(4):759-65. doi: 10.1016/S0022-5223(99)70297-7. PMID 10096972
- [Background] Yellin A, Simansky DA, Paley M, Refaely Y. Hyperthermic pleural perfusion with cisplatin: early clinical experience. Cancer. 2001 Oct 15;92(8):2197-203. doi: 10.1002/1097-0142(20011015)92:83.0.co;2-f. PMID 11596038
- [Background] Iyoda A, Yusa T, Hiroshima K, Fujisawa T. Surgical resection combined with intrathoracic hyperthermic perfusion for thymic carcinoma with an intrathoracic disseminated lesion: a case report. Anticancer Res. 1999 Jan-Feb;19(1B):699-702. PMID 10216479
- [Background] Refaely Y, Simansky DA, Paley M, Gottfried M, Yellin A. Resection and perfusion thermochemotherapy: a new approach for the treatment of thymic malignancies with pleural spread. Ann Thorac Surg. 2001 Aug;72(2):366-70. doi: 10.1016/s0003-4975(01)02786-2. PMID 11515868